CLINICAL TRIAL: NCT04018963
Title: Numerical Simulation Analysis of Nasal Physiology After Endoscopic Pituitary Surgery.
Brief Title: The Impact of Endoscopic Pituitary Surgery on Nasal Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhebao Wu (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor-Investigator, Zhebao Wu, Professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: NSPA-2019
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Pituitary Tumor; Endoscopic Surgery; Quality of Life; Function of Nose
Keywords: Pituitary tumor; Neuroendoscope; Surgical approach; Computational Fluid Dynamics; Numerical simulation
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uninostril group: Subjects will be treated with endoscopic transsphenoidal pituitary surgery with the single nostril approach.
  Interventions: Procedure: Single nostril approach endoscopic transsphenoidal pituitary surgery
- Binostril group: Subjects will be treated with endoscopic transsphenoidal pituitary surgery with the bilateral nostril approach.
  Interventions: Procedure: Bilateral nostril approach endoscopic transsphenoidal pituitary surgery

INTERVENTIONS:
Procedure: Single nostril approach endoscopic transsphenoidal pituitary surgery — Single nostril approach endoscopic transsphenoidal pituitary surgery
  Groups: Uninostril group
Procedure: Bilateral nostril approach endoscopic transsphenoidal pituitary surgery — Bilateral nostril approach endoscopic transsphenoidal pituitary surgery
  Groups: Binostril group

SUMMARY:
The aim of this study is to determine the impact of endoscopic transsphenoidal pituitary surgery on nasal function using a numerical simulation and to compare the difference between two kinds of transsphenoidal approachese(single nostril approach and bilateral nostril approach)．

DETAILED DESCRIPTION:
Neuroendoscopic surgery is the first treatment for most pituitary adenoma patients. Because transsphenoidal surgery exploits the nasal corridor and paranasal sinuses to reach the skull base, sinonasal trauma is a primary source of postoperative morbidity in many of these patients. The aim of this study is to determine the impact of endoscopic transsphenoidal pituitary surgery on nasal function using a numerical simulation and to compare the difference between two kinds of transsphenoidal approachese(single nostril approach and bilateral nostril approach)．

ELIGIBILITY:
Inclusion Criteria:

1. Enhanced MRI shows a pituitary tumor
2. Endoscopic surgery is required according to the pituitary tumor treatment guidelines.
3. Karnofsky performance status ≥ 70.
4. The patient has signed the informed consent.

Exclusion Criteria:

1. Patients who have undergone previous transsphenoidal surgery or other nasal surgery.
2. Patients who had a history of nasal tumors.
3. Patients who had a history of severe head or face trauma.
4. Patients with congenital sinus malformation.
5. Pregnant or lactating women.
6. Patients with serious systemic diseases without control.
7. Patients with poor compliance, who cannot implement the program strictly.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with endoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Nasal airway patency. | Up to 3 months
  A bilateral model of the human nose on a CT-scan will be reconstructed to display geometric parameters of nasal cavity 3 months after surgery.
Airflow patterns. | Up to 3 months
  A bilateral model of the human nose on a CT-scan will be reconstructed. A numerical simulation applying the computational fluid dynamics (CFD) will be performed displaying intranasal airflow patterns 3 months after surgery.
Temperature parameter. | Up to 3 months
  A bilateral model of the human nose on a CT-scan will be reconstructed. A numerical simulation applying the computational fluid dynamics (CFD) will be performed displaying intranasal temperature parameter 3 months after surgery.
Humidity parameter. | Up to 3 months
  A bilateral model of the human nose on a CT-scan will be reconstructed. A numerical simulation applying the computational fluid dynamics (CFD) will be performed displaying intranasal humidity parameter 3 months after surgery.
VAS | Up to 3 months
  Record the Visual Analogue Scale(VAS) 3 months after surgery. The VAS scale includes six sub-scales: rhinorrhea VAS, rhinobyon VAS，rhinocnesmus VAS, cough VAS, sneezing VAS and olfaction VAS. Each scale has a maximum score of 10 and a minimum score of 0. The total VAS was the average of all sub-scales. Higher values represent a better outcome.
CT Lund-Mackay Score | Up to 3 months
  Record the CT Lund-Mackay Score 3 months after surgery.The CT Lund-Mackay Score has a maximum score of 24 and a minimum score of 0. Higher values represent a worse outcome.
SNOT-20 | Up to 3 months
  Record the Sino-Nasal Outcome Record the Test-20(SNOT-20) 3 months after surgery. The SNOT-20 has a maximum score of 60 and a minimum score of 0. Higher values represent a worse outcome.
SF-36 | Up to 3 months
  Record the Medical Outcome Study Short Form 36-items Health survey(SF-36) 3 months after surgery. The SF-36 includes six sub-scales: General Health, Reported Health Transition，Physical Functioning, Role-Physical, Role-Emotional, Social Functioning, Bodily Pain, Vitality and Mental Health. Each scale has a maximum score of 100 and a minimum score of 0. The total score was the average of all sub-scales. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Change on Tumor | Up to 3 months
  Record the tumor volume from enhanced pituitary MRI 3 months after surgery.
Nasal airway patency. | 1 week after surgery
  A bilateral model of the human nose on a CT-scan will be reconstructed to display geometric parameters of nasal cavity 1 week after surgery.
Airflow patterns. | 1 week after surgery
  A bilateral model of the human nose on a CT-scan will be reconstructed. A numerical simulation applying the computational fluid dynamics (CFD) will be performed displaying intranasal airflow patterns 1 week after surgery.
Temperature parameter. | 1 week after surgery
  A bilateral model of the human nose on a CT-scan will be reconstructed. A numerical simulation applying the computational fluid dynamics (CFD) will be performed displaying intranasal temperature parameter 1 week after surgery.
Humidity parameter. | 1 week after surgery
  A bilateral model of the human nose on a CT-scan will be reconstructed. A numerical simulation applying the computational fluid dynamics (CFD) will be performed displaying intranasal humidity parameter 1 week after surgery.
SF-36 | 1 week after surgery
  Record the Medical Outcome Study Short Form 36-items Health survey(SF-36) 1 week after surgery. The SF-36 includes six sub-scales: General Health, Reported Health Transition，Physical Functioning, Role-Physical, Role-Emotional, Social Functioning, Bodily Pain, Vitality and Mental Health. Each scale has a maximum score of 100 and a minimum score of 0. The total score was the average of all sub-scales. Higher values represent a better outcome.
SNOT-20 | 1 week after surgery
  Record the Sino-Nasal Outcome Record the Test-20(SNOT-20) 1 week after surgery. The SNOT-20 has a maximum score of 60 and a minimum score of 0. Higher values represent a worse outcome.
CT Lund-Mackay Score | 1 week after surgery
  Record the CT Lund-Mackay Score 1 week after surgery. The CT Lund-Mackay Score has a maximum score of 24 and a minimum score of 0. Higher values represent a worse outcome.
VAS | 1 week after surgery
  Record the Visual Analogue Scale(VAS) 1 week after surgery. The VAS scale includes six sub-scales: rhinorrhea VAS, rhinobyon VAS，rhinocnesmus VAS, cough VAS, sneezing VAS and olfaction VAS. Each scale has a maximum score of 10 and a minimum score of 0. The total VAS was the average of all sub-scales. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhebao Wu, phd, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Little AS, Kelly D, Milligan J, Griffiths C, Prevedello DM, Carrau RL, Rosseau G, Barkhoudarian G, Otto BA, Jahnke H, Chaloner C, Jelinek KL, Chapple K, White WL. Predictors of sinonasal quality of life and nasal morbidity after fully endoscopic transsphenoidal surgery. J Neurosurg. 2015 Jun;122(6):1458-65. doi: 10.3171/2014.10.JNS141624. Epub 2015 Apr 3. PMID 25839931
- [Background] Tian L, Shang Y, Chen R, Bai R, Chen C, Inthavong K, Tu J. Correlation of regional deposition dosage for inhaled nanoparticles in human and rat olfactory. Part Fibre Toxicol. 2019 Jan 25;16(1):6. doi: 10.1186/s12989-019-0290-8. PMID 30683122
- [Background] McCoul ED, Bedrosian JC, Akselrod O, Anand VK, Schwartz TH. Preservation of multidimensional quality of life after endoscopic pituitary adenoma resection. J Neurosurg. 2015 Sep;123(3):813-20. doi: 10.3171/2014.11.JNS14559. Epub 2015 Jun 5. PMID 26047408